CLINICAL TRIAL: NCT02849366
Title: Combination of Cryosurgery and NK Immunotherapy for Recurrent Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-sarcoma
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma
Keywords: Sarcoma; Cryosurgery; NK Immunotherapy
MeSH Terms: conditions — Sarcoma | interventions — Cryosurgery

ARMS (2):
- Cryosurgery and NK immunotherapy (Experimental): In this group, the patients will receive comprehensive cryosurgery to clear all big tumors and then receive multiple NK immunotherapies. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Cryosurgery; Biological: NK immunotherapy
- Cryosurgery (Active Comparator): In this group, the patients will receive comprehensive cryosurgery to clear all big tumors. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Cryosurgery

INTERVENTIONS:
Device: Cryosurgery — Percutaneous ablation under CT or ultrasound guidance
  Other Names: Argon-helium cryosurgical system
Biological: NK immunotherapy — Each treatment: 8-10 billion cells in all, transfuion in 3 times, i.v.
  Arms: Cryosurgery and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of cryosurgery plus NK immunotherapy to recurrent sarcoma.

DETAILED DESCRIPTION:
By enrolling patients with recurrent sarcoma adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using cryosurgery and natural killer (NK) cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Relief degree | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, MD, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Fuda cancer institute of Fuda cancer hospital, Guangzhou, Guangdong, China